CLINICAL TRIAL: NCT06976554
Title: Mechanical Ventilator Weaning in Chronically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Barlow Respiratory Hospital (Unknown)
Responsible Party: Principal Investigator, Tamas Dolinay, MD, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-001420
Record Dates: First submitted 2025-04-28; First posted 2025-05-16 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Mechanical Ventilation Complication
Keywords: prolonged mechanical ventilation; ventilator weaning; tracheostomy
MeSH Terms: interventions — Weaning

STUDY DESIGN:
Intervention Model Description: Randomized to intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapist-implemented patient-specific (TIPS) ventilator weaning (Active Comparator): In the TIPS path, participants will complete a 21 step protocol. Mechanical ventilator (MV) weaning is done with synchronized intermittent mandatory ventilation (SIMV) mode for 24 hrs. Patients will transition to this mode on the Day 1 (D1) after completion of SBT. The initial ventilator setup is PS 20 cmH2O PEEP 5cmH2O set RR 10/min. During the first 4 steps the backup rate will be lowered gradually from 8/min to 4/min (Step 1-4). Subsequently the PS will be reduced from 20 to 10 by each step (Step 5-9). SBT is performed in Step 10 with 1 hr. CA trials. ABG is performed in Step 11 with 2 hrs. of CA to assure respiratory stability. Patients rest on SIMV PS=10 cmH2O PEEP=5cmH2O, RR=4 (Step 9) setting during CA trial. Subjects can progress up to 3 steps daily, if deemed able by the respiratory therapist. The protocol completes when the patients is able to complete 72 hours of continuous CA time.
  Interventions: Procedure: weaning
- Pressure support ventilation (PSV) weaning (Active Comparator): In the PSV path, participants will complete a 14-step protocol. In this protocol gradual decrease of PS is used for 10-12 hrs. a day. PS is decreased from 20cmH2O to 10cmH2O with 5cmH2O PEEP applied (Step 1-6). Every weaning step is followed by rest on the same ventilator setting the patient had on admission. Starting Step 7, subjects will undergo daily SBT (1 hour 5cmH2O PS with 5cmH2O PEEP). If they pass, they will progress to CA trials (Step 8-14). ABG is performed after 2 hours of CA time in Step 7 to assure respiratory stability. CA time will be extended by 4 hrs. in Step 8 to 14. Patients rest on the admission ventilator settings. Subjects can progress up to 3 steps daily, if deemed able by the respiratory therapist. The protocol completes when the patients is able to complete 72 hrs. of continuous CA time.
  Interventions: Procedure: weaning

INTERVENTIONS:
Procedure: weaning — gradual weaning from the mechanical ventilator

SUMMARY:
Mechanical ventilation is a commonly used life-saving hospital procedure for patients with severe breathing difficulty. Some patients have difficulty separating from the ventilator and need to be removed gradually. This process is called ventilator weaning. It is not known what is the best way to wean patients from the ventilator. In this study, the investigators will compare two commonly used ventilator weaning strategies and compare their success. One ventilator strategy, the Pressure Support Ventilation weaning (PSV), combines 12 hours ventilator weaning with 12 hours rest on the ventilator. This strategy is faster with an anticipated weaning in 2 weeks. The other strategy, the Therapist implemented Patient Specific weaning (TIPS), gradually lowers support and weans in 3 weeks.

Patients admitted to Barlow Respiratory Hospital (BRH) for ventilator weaning will be asked to participate in this study within 72 hours of hospital admission. Participants will undergo a spontaneous breathing trial (SBT) to assess your ability to breathe while receiving minimal or no ventilator support. Patients who pass SBT will be eligible for cool aerosol trials (humidified, oxygenated air without positive pressure mechanical ventilation). Participants who fail SBT within 24 hours will be eligible for the study. Participants will be randomized to receive PSV or TIPS ventilator weaning. The investigators will collect clinical, laboratory and mechanical ventilator information throughout the study period. Ventilator weaning success will be compared at day 30. The study will not interfere with any components of clinical care but the study investigators will be allowed to change the ventilator weaning strategy from PSV to TIPS, if a participant is unable to tolerate PSV weaning.

DETAILED DESCRIPTION:
Study protocol:

1. Patients will be considered for enrollment in the study within 72 hours of admission to BRH.
2. All Barlow Respiratory Hospital (BRH) patients requiring positive pressure invasive mechanical ventilation (MV) undergo spontaneous breathing trial (SBT, pressure support ventilation (PS) 5cmH2O with 5cmH2O of positive end expiratory pressure, PEEP) per hospital policy within 24 hours of admission. Patients who pass SBT will be eligible for cool aerosol trials (humidified, oxygenated air without positive pressure mechanical ventilation). These patients will be excluded from the study, except if a patient fails to tolerate cool aerosol within 24 hours and continue require continuous positive pressure ventilation. These patients can be considered for study enrollment the next day.
3. In the rare instance that a patient has an endotracheal tube on admission to BRH and continued MV is needed, a date for tracheostomy will be set. Patients following tracheostomy placement can participate in the study.
4. Parameters to preclude study enrollment are listed in the Exclusion criteria.
5. All patients are admitted to monitored beds at BRH. Vital signs (heart rate, oxygen saturation and lead 2 electrocardiogram, respiratory rate and ventilator compliance) are continuously monitored. Blood pressure is measured every 6 hours. Hemodynamic and respiratory stability is assessed daily on these parameters by the nurse and the respiratory therapist.
6. On the first day of the study, Day0 (D0), if a patient is stable and required continued MV, the study team will approach the patient and/or the patient's designated power of attorney (DPOA) for informed consent.
7. On D0, consented patients, now referred to as participants, will be randomized to participate in PSV or TIPS ventilator weaning.
8. On Day 1 (D1), weaning starts. Hemodynamic and respiratory instability is assessed every day as in point 5. Unstable participants will complete the study, but will be followed throughout their hospitalization at BRH for hospital outcomes. Further weaning can be attempted after stabilization outside of the study protocol per the hospital weaning program.
9. If a participant fails to progress to the next step of ventilator weaning, the same step can be repeated on 3 consecutive days and if possible can continue with the designated weaning path.
10. If a participant cannot progress beyond the same step after 3 consecutive days in the PSV path, the participant will continue with TIPS path step 1.
11. If a participant cannot progress beyond the same step after 3 consecutive days in the TIPS path, the participant will complete the study.
12. Both paths will consist of a MV and a cool aerosol (CA) trial parts. The length of the TIPS path is a minimum 21 steps and 14 steps for the PSV path. These usually refer to days, but subjects may progress up to 3 steps in a day. The details of both path are shown in the "ventilator paths" section.
13. When a participant is transitioned from MV to CA, arterial blood gas (ABG), will be collected after 2hrs CA to ensure adequate oxygenation and to avoid elevated carbon dioxide levels.
14. Following completion of the study all participants will be assessed for tracheostomy decannulation by pulmonology, speech pathology and respiratory therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients requiring positive pressure mechanical ventilation for at least 21 days prior to BRH admission and
2. Have a secure tracheostomy.

Exclusion Criteria:

1. Inability to obtain informed consent from patient or DPOA
2. Incarcerated patients
3. Patients with less than 3 months of life expectancy
4. Patients requiring vasopressor medication to stabilize blood pressure on admission
5. Systolic blood pressure less than 90mmHg on admission
6. Pulse less than 50 or greater than 130 beats per minute or change by more than 20 from baseline on admission
7. Respiratory rate greater than 35/min
8. Oxygen saturation less than 90%
9. PEEP>5cmH2O
10. Lung tidal volume less than 250ml despite MV support
11. At least one previous admission to BRH with unsuccessful ventilator liberation attempt
12. Length of Stay (LOS) at BRH less than 24hours
13. Patients pass spontaneous breathing trial (SBT) on D1 and eligible for cool aerosol, except if they fail SBT on D2 and require continued MV

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
weaning success | 30 days
  Patients who can disconnect from the mechanical ventilator for 3 consecutive days or have their tracheostomy decannulated will be considered weaned ("success") and will have completed the protocol.

SECONDARY OUTCOMES:
tracheostomy decannulation | 30 days
  Tracheostomy decannulation
hospital length of stay | throughout study completion, an average 90 days
  Hospital length of stay
intensive care unit admissions | 30 days
  Intensive care unit admissions at Barlow Respiratory Hospital
in-hospital mortality | throughout study completion, an average 90 days
  In-hospital mortality at Barlow Respiratory Hospital
physical activity score | throughout study completion, an average 90 days
  Physical activity score on admission and at discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Barlow Respiratory Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Only deidentified data will be shared with the study team. This includes health demographics, comorbidities, blood laboratory values, vital signs, ventilator parameters, antibiotics, vasopressors use, health outcomes and discharge location.